CLINICAL TRIAL: NCT03087461
Title: Bridging the Gap: Incorporating Exercise Evidence Into Clinical Practice in Breast Cancer Care in Ontario
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Jenna Smith, PhD Candidate, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HamiltonHSC-JS
Record Dates: First submitted 2017-03-07; First posted 2017-03-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise; Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive a multi-component KT intervention. This will include exercise and self-management components.
  The exercise intervention will involve a moderate intensity aerobic exercise program, using recumbent bikes, delivered within the cancer institution. Participants will take part in the 30-minute sessions 8 times. The intervention will be supervised by a physiotherapist (PT) educated in cancer rehabilitation.
  The SM component will include educational modules created by a PT. Participants will view these 30 minute modules prior to each exercise intervention, over the same 8 sessions.
  Interventions: Behavioral: Exercise and self-management
- Usual Care (No Intervention): Control group receiving usual care (no exercise or self-management education within the institution).

INTERVENTIONS:
Behavioral: Exercise and self-management — The intervention will include aerobic exercise and self-management education using technology.
  Arms: Intervention Group

SUMMARY:
Breast cancer (BC) and its treatments lead to numerous side effects that affect a person's life for years after treatment has ended. Research shows that regular exercise limits many of these side effects. However, less than 30% of BC survivors regularly exercise due to many barriers that include patients being unaware of the benefits of exercise, health professionals facing institutional, personal, and patient-related barriers to promoting exercise, and a lack of knowledge translation (KT) strategies within cancer institutions that focus on accessible exercise interventions and education by physiotherapists. For this project, a pilot study is needed as the first step in order to assess process and resource variables before implementation of a large-scale intervention.

The primary objective of this pilot trial is to assess the feasibility of conducting a larger trial to evaluate the effects of a novel KT intervention using exercise and self-management versus usual care among BC survivors. The secondary objective is to determine preliminary estimates of effects of the KT intervention of exercise plus self-management (SM) program versus usual care on (a) levels of exercise knowledge and behaviour, (b) health related quality of life and (c) resource utilization, among BC survivors over a four month period.

DETAILED DESCRIPTION:
Study Design: Pilot randomized controlled trial. Eligibility: Women older than 18 years who are currently undergoing chemotherapy treatment for BC.

Intervention: The intervention group includes an 8-session multi-component intervention with a structured aerobic exercise program plus SM supervised by a physiotherapist.

Setting: Outpatient-Juravinski Cancer Centre in Hamilton, ON. Control: Usual care. Randomization: Participants will be randomly allocated using a 1:1 allocation ratio to receive the intervention of structured exercise plus SM program or usual care.

Sample size: The study will recruit n=12 number of participants/group for a total of 24 in both groups.

Analysis: A blinded assessor will assess outcomes at baseline, post intervention, at 2- and 4-month follow up. Intervention feasibility and effectiveness will be assessed using descriptive statistics and analysis of covariance for continuous outcomes.

Anticipated Impact: This study aims to assess the feasibility of a larger trial to determine effective ways to close the current KT gap and increase exercise awareness for women with BC. This project will assess process and resource variables before implementation of a larger scale intervention. Together, the overall project goal is to promote sustainable exercise behaviour to help manage the burden of BC.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling, English-speaking women, over 18 years, who are currently undergoing chemotherapy for Stage 1-3 BC and have been cleared by their oncologist to participate in moderate intensity aerobic exercise

Exclusion Criteria:

* Participants will be excluded from the study if they have another chronic disease, cognitive impairment or injury that prevents them from participating independently in moderate intensity exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Study Recruitment Rate: percentage of eligible patients recruited | Baseline
  A recruitment log will be kept, detailing reasons for non-participation.
Intervention Retention Rate: percentage of consented participants who completed the intervention | Post-intervention (2 months post baseline)
  Attendance will be tracked on the feasibility data collection sheet and reasons for non-participation on scheduled intervention days will be documented using an adherence log
Intervention Adherence Rate: percentage of total intervention sessions attended | Post-intervention (2 months post baseline)
  Attendance will be tracked on the feasibility data collection sheet and reasons for non-participation on scheduled intervention days will be documented using an adherence log

SECONDARY OUTCOMES:
Health related quality of life | Baseline, post intervention (2 months post baseline), 2 and 4 month follow up (post intervention completion)
  Functional Assessment of Cancer Therapy-Breast
Exercise knowledge | Baseline, post intervention (2 months post baseline), 2 and 4 month follow up (post intervention completion)
  Theory of planned behaviour questionnaire
Exercise behaviour | Baseline, post intervention (2 months post baseline), 2 and 4 month follow up (post intervention completion)
  Theory of planned behaviour questionnaire
Health status | Baseline, post intervention (2 months post baseline), 2 and 4 month follow up (post intervention completion)
  European Quality of Life-Five Dimension (EQ-5D)
Use of health care services | Baseline, post intervention (2 months post baseline), 2 and 4 month follow up (post intervention completion)
  Piloted form assessing doctor visits, procedures, medication use, missed days of work
Physical Activity Level | Baseline, post intervention, 2 and 4 month follow up
  Godin Leisure Time Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Smith-Turchyn, PT, PhD(c), Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith-Turchyn J, Richardson J, Tozer R, McNeely M, Thabane L. Bridging the gap: incorporating exercise evidence into clinical practice in breast cancer care. Support Care Cancer. 2020 Feb;28(2):897-905. doi: 10.1007/s00520-019-04897-9. Epub 2019 Jun 5. PMID 31168711